CLINICAL TRIAL: NCT06131203
Title: Performance Evaluation of the DeepView AI-Burn For Assessment of Thermal Burn Healing Potential
Brief Title: Burn Validation Study
Acronym: BVS
Status: Completed | Type: Observational
Sponsor: SpectralMD (Industry)
Responsible Party: Sponsor
Other Study IDs: CLA-PR-01
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Burns; Wound Heal; Wounds and Injuries
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Emergency Department Burn Subjects: Subjects with Thermal Burn Injury enrolled through the emergency department
  Interventions: Device: DeepView SnapShot Portable (DV-SSP)
- Burn Center Burn Subjects: Subjects with Thermal Burn Injury enrolled through the burn center
  Interventions: Device: DeepView SnapShot Portable (DV-SSP)

INTERVENTIONS:
Device: DeepView SnapShot Portable (DV-SSP) — DV-SSP assistive imaging to collect observational data

SUMMARY:
The purpose of this study is to validate the algorithm for burn healing assessment by the Spectral MD DeepView device which would provide burn healing potential assessment.

ELIGIBILITY:
Inclusion Criteria:

Willing and able to give informed consent or have a Legally Authorized Representative (LAR) able to do so; Life expectancy > 6 months; Thermal burn mechanism (flame, scald, or contact); The Study Burn(s) occurred less than 72 hours prior to the time of first imaging; and Minimum burn wound size for adult or pediatric patients is 0.5% TBSA per region For adult Subjects: Have 2 - 4 regions of their clinical burn(s) that meet the criteria for a Study Burn.

For pediatric Subjects: Have 1 - 4 regions of their clinical burn(s) that meet the criteria for a Study Burn

Exclusion Criteria:

Burn pattern distribution isolated to head, face, neck, hands, feet, genitalia, and/or joints; Subject has burns involving > 50% total body surface area (TBSA); Sepsis at the time of enrollment; Immunosuppression/radiation/chemotherapy < 3 months prior to enrollment; Concurrent use of investigational products with a known effect on the burn sites; and/or Any condition that in the opinion of the Investigator may prevent compliance with the study requirements or compromise subject safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects enrolled in this study will be recruited at the designated Study Site within 72 hours of suffering a thermal burn injury. Adult and pediatric Subjects with burns from one or more of the defined burn severities will be enrolled. All Subjects must meet the specified inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Primary BC Endpoint | 3 weeks
  Demonstrate the DeepView AI-Burns' sensitivity is superior to BC HCPs' bedside examination while maintaining non-inferior specificity to burn HCPs.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Valleywise Health, Phoenix, Arizona
  - Shriners Children's Northern California, Sacramento, California
  - University of California Davis Health, Sacramento, California
  - University of California San Diego, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook Medical Center, Stony Brook, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Ohio State University, Columbus, Ohio
  - St. Christopher's Children Hospital, Philadelphia, Pennsylvania
  - MUSC Shawn Jenkins Children's Hospital, Charelston, South Carolina
  - Texas Tech University, Lubbock, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Harborview, Seattle, Washington